CLINICAL TRIAL: NCT06591000
Title: Clinical Efficacy and Long-term Outcomes of Allograft Versus Stented Biological Prosthesis for Primary Tricuspid Valve Disease
Brief Title: Clinical Efficacy and Long-term Outcomes of ALLOgraft Versus Stented Biological Prosthesis for Primary TRIcuspid Valve Disease (ALLOTRI)
Status: Recruiting | Type: Observational
Sponsor: Chelyabinsk Regional Clinical Hospital (Other Government)
Responsible Party: Principal Investigator, Mikhail Nuzhdin, Director, Chelyabinsk Regional Clinical Hospital
Other Study IDs: 14012016
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Allograft; Bioprosthesis; Tricuspid Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allograft tricuspid valve replacement: Patients underwent mitral allograft implantation for primary tricuspid valve disease
  Interventions: Procedure: tricuspid valve replacement
- Stented biological tricuspid valve replacement: Patients underwent biological stented valve replacement for primary tricuspid valve disease
  Interventions: Procedure: tricuspid valve replacement

INTERVENTIONS:
Procedure: tricuspid valve replacement — Complete or partial tricuspid valve replacement with mitral allograft/ complete tricuspid valve replacement with biological prosthesis

SUMMARY:
The aim of the study is to evaluate early safety, clinical efficacy and long-term outcomes of mitral allografts and stented biological prosthesis in tricuspid valve replacement for primary tricuspid valve diseases.

DETAILED DESCRIPTION:
Early safety (morbidity, mortality rate, freedom from any valve related complication) along with clinical efficacy ( survival, freedom from reoperation, repeat endocarditis and other valve related complication ), long term outcomes ( survival, freedom from reoperation, repeat endocarditis and other valve related complication ), echocardiografic assessment and MSCT scan for both groups of patients are going to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary tricuspid valve disease and/or tricuspid bioprosthetic failure scheduled for tricuspid valve intervention.

  * Intraoperative findings suggested for tricuspid valve replacement rather than repair.

Exclusion Criteria:

* Pregnancy

  * Confirmed active drug addiction
  * Progressive HIV-infection
  * HIV-infected patients with CD4-cells count less than 250
  * Patients with secondary tricuspid valve pathology (left-sided valve disease)
  * LV Ejection fraction less than 40%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary tricuspid valve disease and/or tricuspid bioprosthetic failure scheduled for tricuspid valve intervention
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2016-01-14 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day period after surgery
  Freedom from all-cause mortality (%)
Stroke | 30-day period after surgery
  Stroke rate (n,%)
Severe valve dysfunction | 1-year after surgery, annually, assessed up to 3 years
  Number of patients free from peak valve gradient more than 6 mmHg and severe valve regurgitation (vena contracta no more than 6 mm), (n,%)
Freedom from prosthetic endocarditis | 1-year after surgery, annually, assessed up to 3 years
  Number of patients free from prosthetic endocarditis (n,%)
Freedom from reoperation | 1-year after surgery, annually, assessed up to 3 years
  Number of patients free from secondary operation due to severe valve (n,%) dysfunction (n,%)
New pacemaker implantation | 1-year after surgery, annually, assessed up to 3 years
  Number of patients, free from pacemaker implantation after surgery (n,%)

SECONDARY OUTCOMES:
Transvalvular gradient | 1 year after surgery, annually, assessed up to 3 years
  Peak and mean gradient (mmHg)
Transprosthetic regurgitation | 1 year after surgery, annually, assessed up to 3 years
  Vena contracta (mm)
Right atrial remodeling | 1 year after surgery, annually, assessed up to 3 years
  right atrium size (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Malinovsky, PhD, Study Chair — Department of Cardiac Surgery
Locations (1):
- Department of Cardiac Surgery, Chelyabinsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nuzhdin M, Malinovsky Y, Galchenko M, Komarov R, Fokin A, Nadtochiy N. Stented Biological Prosthesis Versus Mitral Allograft in Surgical Treatment of Tricuspid Valve Infective Endocarditis. Rev Cardiovasc Med. 2025 Jul 8;26(7):37204. doi: 10.31083/RCM37204. eCollection 2025 Jul. PMID 40776959